CLINICAL TRIAL: NCT04788121
Title: Efficacy of Early Administration of Tranexamic Acid in Upper Gastrointestinal Bleeding: A Randomized Controlled Trial
Brief Title: Efficacy of Tranexamic Acid in Upper Gastrointestinal Bleeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGI/IEC/2020/001466
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Gastro Intestinal Bleeding
Keywords: GI bleed, Tranexamic Acid
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Tranexamic Acid; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment/Tranexamic Acid Group (Active Comparator): The treatment group will receive Injection TXA 1gm intravenous (IV) over 15 minutes infusion dissolved in 100 ml normal saline (NS- 0.9% NaCl), followed by injection TXA 2 g IV over 12 hours infusion dissolved in a 500 ml NS.
  Interventions: Drug: Tranexamic acid; Other: Standard of care
- Control Group (Placebo Comparator): The control group will receive injection 100 ml NS over 15 minutes infusion, followed by injection 500 ml NS over 12 hours infusion.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Tranexamic acid — The treatment group will receive Injection TXA 1gm intravenous (IV) over 15 minutes infusion dissolved in 100 ml normal saline (NS- 0.9% NaCl), followed by injection TXA 2 g IV over 12 hours infusion dissolved in a 500 ml NS
  Arms: Treatment/Tranexamic Acid Group
Other: Standard of care — For management, initial priority will be given to secure airway, breathing and circulation. To ensure hemodynamic stability, crystalloids infusion will be given as and when required. Blood transfusion will be initiated at the threshold hemoglobin (Hb) of 7g/dl, to maintain the target Hb of 7-9g/dl or with signs of hemodynamic instability despite fluid resuscitation. Intra venous (IV) PPI and antibiotic will be started promptly in all cases and IV splanchnic vasoconstrictor will be given in all suspicious case of Variceal hemorrhage before definitive therapeutic and diagnostic endoscopic procedure is done.

SUMMARY:
Upper Gastrointestinal bleed is a common presentation in a medical emergency. Patients generally present with hematemesis, melena or in severe cases hematochezia. Incidence and etiology vary from region as well as the level of health care facility. In the US, UGI bleed accountsfor about 300000 admissions per year (6). India has a huge burden of UGI bleed. A study in India showed 4.6% of hospitaladmissions were due to UGI bleed (7). As per the medical record of PGIMER, 2-3 patients of UGIbleed are admitted to the EMOPD every day.

Upper GI bleed is anatomically defined as any gastrointestinal bleed originating proximal to ligamentof treitz (8). Causes of UGI bleed are generally divided into variceal and non-variceal in origin. The common etiology of non-variceal bleed are Peptic Ulcer disease (PUD), esophagitis, erosive Gastritis, vascular malformations, Mallory Weiss tear and GI malignancies.Variceal hemorrhage is usually secondary to esophageal varices, but alsocan be due to gastric varices and ectopic varices of the upper GI tract(9).Non-varicealcauses are more common as compared to variceal bleed (10) and among this PUD is the most common (10).But there is recent rising trend of variceal bleed secondary to chronic liver disease and portal hypertension .As per a recently published institutional study, variceal bleed constituted 45.7% of UGI bleed (11). Morbidity and mortality associated with UGI bleed are significantly high.Variceal bleed is becoming a major concern in tertiarycare centers and carries a higher mortality as compared to non variceal bleed(12 ).Clinical severity of UGI bleed may vary from being insignificant to fatal. Mortality from UGI bleed may vary from 2 to 5% where as it around 10-30% in cases of re-bleed (12). Prompt UGI endoscopic procedure is diagnostic as well as therapeutic which should be done ideally within first 24hrsalong with airway, volume and blood resuscitative measures (13).High dose proton pump inhibitors(PPI) are used for non-variceal bleed where as splanchnic vasoconstrictorsare used in variceal bleed along with endoscopic procedure like injection of Epinephrine, Sclerosants, application of haemostatic material like hemoclips/endoclips, over the scope clips, glue or tissue adhesive, haemostatic powder/spray. Beside these endoscopic bipolar electro coagulation, heater probe coagulation, argon plasma coagulator, laser photocoagulation can also be done as and when required. For variceal bleed endoscopic variceal band ligation (EVL) is the main stay of therapy. However routine use of antifibrinolytic agent hasn't been recommended in the guidelines for management of acute UGI bleed.

Studies have shown that fibrinolysis may play an important role in GI bleeding dueto premature breakdown of fibrin blood clots at the bleeding site (14). Studies have also shown that many patients with acute UGI bleed have elevated levels of fibrin degradation products (a surrogate marker for fibrinolysis) and that is associated with worse outcomes (14). Fibrinolysisalso contributes to the risk of re-bleed.Literature review suggests that early administration ofTranexamic acid (TXA) reduces mortality due to bleeding in trauma patients (15) and effective in controlling bleeding in menorrhagia (16). Our own institutional study showed that TXA is effective as a bridging therapy in controlling bleeding from haemoptysis before definitive therapeutic intervention done (1). A systematic COCHRANE review of TXA in UGI bleed identified 7 trials (3). These trials showed statistically significant reduction in mortality and reduced need ofsurgical interventions in patients receiving TXA. However the trials had many fallacieslike small sample size, number of biases. The NICE guideline doesn't include TXA inthe management of GI bleed (4). So far studies on use of TXA in UGI bleed haven't been able to either recommend or refute the use of TXA in UGI bleed (3).

There is also lack of study form India and the Southeast Asia regarding the efficacy of TXA in UGI bleed. TXA, an anti-fibrinolytic agent, inhibits fibrinolysis by displacing plasminogen from fibrin. So, TXA may have role in bleeding control and preventing re-bleed in acute UGI bleed by stabilization of the clot formation. This study will evaluate the efficacy of early administration of TXA in acute onset UGIbleed, in term of bleeding control, preventing re-bleeding and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Irrespective of gender and with age ≥ 18 years, all the patients presenting with symptoms of acute UGI bleed will be enrolled for the study after taking written informed consent.

Exclusion Criteria:

1. Patients with UGI bleed for more than 48 hours, history of UGI bleed in previous 1 year
2. Chronic kidney disease
3. Pregnancy and breast feeding
4. Malignancy
5. Patients who have already received TXA
6. UGI endoscopy done beyond 24 hours of admission because of hemodynamic instability or encephalopathy
7. Patients who will be receiving blood thinners like anti-platelets, anti-coagulation agents within 4 weeks of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding control | 24 hours
  Bleeding control is defined as:
  1. No active hematemesis or no blood in the nasogastric (NG) aspirate (100 ml) > 2hrs after start of standard treatment.
  2. Absence of persistent shock or absence of installation of shock after initial contact (SBP<90/MAP<60/HR>100/min).
  3. No introduction or no increase of systemic vasopressors (except Terlipressin).
  4. Hemoglobin drop < 3gm/dl from the baseline within any 24 hour period if no transfusion is administered.
Re-bleed | 72 hours
  Re-bleed is defined as:
  1. Hb drop of >2g/dl after 2 consecutive stable values > 3hours apart.
  2. Persistently dropping Hb>3g/dl in 24 hours associated with persistent hematemesis or malena.
  3. Development of new onset tachycardia (HR>110/min) or hypotension (SBP<90) after >1 hour of hemodynamic stability.
  4. New onset overt hematemesis.
  5. Presence of bright red blood in the stomach or duodenum or both at repeat endoscopy when more bleeding was suspected.

SECONDARY OUTCOMES:
Mortality | 4 weeks
  incidence of death
Change in D-dimer level | 24 hours
  Change in D-dimer level before and after TXA therapy
ADR | 24 hours
  Incidence of adverse drug reaction
Duration of hospital stay | 4 weeks
  Duration of hospital stay in numbers of days
Need for blood transfusion | 72 hours
  Number of Packed red blood cell (PRBC) need to be transfused

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is available with the principal investigator which may be considered for availability to others as per institutional ethic committee direction.